CLINICAL TRIAL: NCT05848024
Title: Prospective, Single-Center, Non-Controlled, Non-Randomized, Open Study Evaluating the Performance and Stability of Amistem® C
Brief Title: EBRA Study AMISTEM-C FR
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.001.10
Record Dates: First submitted 2023-04-21; First posted 2023-05-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Primary objective: Evaluate femoral stem migration Secondary objective: Evaluate the performance of AMIStem H Proximal Coating at 10 years after surgery; assessment of functional recovery; radiological evaluation; reporting of complications

Scores collected:

HHS, OHS, PMA, UCLA

DETAILED DESCRIPTION:
The main objective of the study was to evaluate the migration and performance of the AMIStem® C femoral stem at 10 years follow-up.

The primary endpoint is the measurement of femoral component migration by EBRA-FCA (The Ein Bild Roentgen Analyse-femoral component analysis, Innsbruck, Austria)

The secondary objectives of the study are:

Evaluate the performance of the AMIStem® C stem Evaluate the function of the operated hip To evaluate the quality of life To evaluate the safety of the AMIStem® C femoral stem Evaluate the postoperative stability and fixation of the hip prosthesis

ELIGIBILITY:
The inclusion criteria are:

1. Patient with a disease (primary coxarthrosis, inflammatory arthritis of the hip, necrosis of the femoral head...) requiring the placement of a total hip prosthesis.
2. Patient who will receive an AMIStem® C cemented femoral stem.
3. Patient willing to comply with the study requirements
4. Patient who has signed the information letter agreeing to the processing of their data in the clinical evaluation
5. Patient affiliated to a social security system
6. Patients aged 18 to 85 years

The criteria for non-inclusion are:

1. Participation in biomedical research
2. Minor patients
3. Protected adult patients
4. Vulnerable persons according to article L1121-6 of the Public Health Code
5. Pregnant or breastfeeding women
6. Patients unable to formulate their non-opposition
7. Patient refusing collection of personal data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a disease (primary coxarthrosis, inflammatory arthritis of the hip, necrosis of the femoral head, etc.) requiring a total hip replacement and who will receive an AMIStem® C cemented femoral stem.
  Patients will be able to participate in other non-interventional research during the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Assess the femoral stem migration | 2 years
  The primary endpoint is the measurement of femoral component migration by EBRA-FCA software (The Ein Bild Roentgen Analyse-femoral component analysis, Innsbruck, Austria) with an accuracy of ± 1.5 mm (95% percentile), a specificity of 100% and a sensitivity of 78% for the detection of a migration of more than 1.0 mm, referring to the RSA method. The EBRA-FCA method is based on the detection of 19 points on the bony femur and the femoral component, as well as two lines to determine the axis of the implant on successive radiographs of the front pelvis. The correction of the radiological enlargement is performed based on the known diameter of the prosthetic femoral component. Lengths are measured from anatomical reference points to ensure comparability of the radiographs. The change in the distance between the top of the greater trochanter and the shoulder of the prosthesis is used to measure the migration of the femoral component.

SECONDARY OUTCOMES:
Assess the AMIStem C performance at 10 years | 10 years
  The survival rate according to a Kaplan Meier curve. The Kaplan-Meier method calculates the survival of the prosthesis by measuring the fraction of living subjects during a period after the procedure. Each time an expected event occurs (revision of the prosthesis, patients lost to follow-up, death, etc.), the probability of implant survival changes. This information is used to estimate the performance of the prosthesis.
  During the study, the number of stem revisions and the number of patients who died or were lost to follow-up will be collected to calculate the probability of survival. The time of occurrence will be recorded for each event.
Assess the functionality of the operated hip | pre-op, 7 days, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Evaluation of the Harris Hip Score The Harris Hip Score (HHS) items include an analysis of the operated hip according to pain, function, mobility, stability and deformity analysis. The Harris Hip Score will be used to assess the patient's subjective and objective improvement in the above criteria. The usefulness of this score has been studied to estimate the clinical results after THR, it is a reference score in the field of orthopedics.
  The Harris hip score is scored from 0 (worst functional outcome and maximum pain) to 100 points (best functional outcome and least pain).
Assess the Quality of Life of patients | pre-op, 7 days, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Merle d'Aubigné functional score The Postel and Merle d'Aubigné (PMA) score: a method for grading the functional value of the hip form a minimum of 0 to a maximum of 18 points.
Assess the security of AMIStem C and collect complications | pre-op, 7 days, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Collection of intra- and postoperative complications (infection, loosening,etc)
Assess the postoperative stability and fixation of AMIStem C | pre-op, 7 days, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Collection of Oxford Hip Score: It is a score composed of 12 questions evaluating the function and pain of the hip before and after arthroplasty.
  The scores for the 0-48 scale can be interpreted as follows[6]:
  Score 0 to 19 May indicate severe hip arthritis. It is highly likely that you may well require some form of surgical intervention, contact your family physician for a consult with an orthopaedic surgeon.
  Score 20 to 29 May indicate moderate to severe hip arthritis. See your family physician for an assessment and x-ray. Consider a consult with an orthopaedic surgeon.
  Score 30 to 39 May indicate mild to moderate hip arthritis. Consider seeing your family physician for an assessment and possible x-ray. You may benefit from non-surgical treatment, such as exercise, weight loss, and/ or anti-inflammatory medication.
  Score 40 to 48 May indicate satisfactory joint function. May not require any formal treatment.
Radiological analysis | pre-op, 7 days, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  -Standard X-ray to identify radiolucencies and endosteal cavitations

CONTACTS AND LOCATIONS:
Overall Officials: Donatien Bocquet, Principal Investigator — Hôpital privé Arras Les Bonnettes 2 rue du docteur Forgeois 62012 Arras
Locations (1):
- Hôpital privé Arras Les Bonnettes, Arras, France

IPD SHARING:
Plan to Share IPD: No